CLINICAL TRIAL: NCT06232148
Title: Procedural Cost Analyses of Robotic Ventral Hernia Repair Compared With Laparoscopic or Open Repair: A Cohort Study
Brief Title: Cost Evaluation of Robotic Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kristian Kiim Jensen, Principal investigator, MD, PhD, DmSci, Bispebjerg Hospital
Other Study IDs: robotic hernia repair
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Ventral Hernia
Keywords: cost
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robotic ventral hernia repairs
  Interventions: Device: Type of surgery
- Open ventral hernia repairs
- Laparoscopic ventral hernia repairs

INTERVENTIONS:
Device: Type of surgery
  Groups: Robotic ventral hernia repairs

SUMMARY:
To evaluate the procedural cost of robotic ventral hernia repair compared with open ventral hernia repair.

DETAILED DESCRIPTION:
Ventral hernia repair is one of the most frequently performed elective surgeries worldwide. The surgical approaches vary depending on the patient characteristics, type, and location the of ventral hernia, as well as the surgeons' preferences and equipment availability.

The choice between an open or minimally invasive approach has been debated for years, and it seems clear that the risk of wound infection is significantly decreased when choosing a minimally invasive approach, whereas there are no significant difference in recurrence rates. In the past decades, the use of a robotic system for ventral hernia repair has gained increasing popularity due to an easy access to the preperitoneal or retromuscular plane with a minimally invasive technique.

Two nationwide cohort studies concluded that length of stay and postoperative morbidity was decreased for robot-assisted repairs compared to open or laparoscopic ventral hernia repairs. Critics of robot-assisted surgery argue that it is time-consuming, too expensive, and that further cost-effectiveness analyses are needed to weigh the clinical benefits.

The aim of these studies was to compare the procedure-specific cost of robot-assisted with open primary ventral and incisional hernia repair and thereafter with laparoscopic repairs.

ELIGIBILITY:
Inclusion Criteria: patients undergoing elective primary ventral and incisional hernia repair -

Exclusion Criteria: none

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing ventral hernia repair in the inclusion period
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Mean procedural cost | at the procedure
  Total mean cost per procedure for all types of ventral hernias

SECONDARY OUTCOMES:
Cost incisional | at the procedure
  Total mean cost per procedure for incisional ventral hernias
Cost primary ventral | at the procedure
  Total mean cost per procedure for primary ventral hernias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henriksen NA, Helgstrand F, Jensen KK. Short-term outcomes after open versus robot-assisted repair of ventral hernias: a nationwide database study. Hernia. 2024 Feb;28(1):233-240. doi: 10.1007/s10029-023-02923-8. Epub 2023 Nov 30. PMID 38036692
- [Background] Jensen KK, Helgstrand F, Henriksen NA. Short-term Outcomes After Laparoscopic IPOM Versus Robot-assisted Retromuscular Repair of Small to Medium Ventral Hernias: A Nationwide Database Study. Ann Surg. 2024 Jan 1;279(1):154-159. doi: 10.1097/SLA.0000000000005915. Epub 2023 May 22. PMID 37212128